CLINICAL TRIAL: NCT03023228
Title: Diabetes To Go: A Pilot Feasibility and Preliminary Efficacy Evaluation of an Inpatient Diabetes Self-management Survival Skills Education Program
Brief Title: Diabetes To Go: An Inpatient Diabetes Survival Skills Education Program
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medstar Health Research Institute (Other)
Collaborators: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 2009-354
Record Dates: First submitted 2015-05-04; First posted 2017-01-18 (Estimated); Last update posted 2020-08-18 (Actual); Status verified 2017-01

CONDITIONS: Diabetes Mellitus; Hyperglycemia
Keywords: Diabetes mellitus; Hyperglycemia; Inpatient; self-management education
MeSH Terms: conditions — Diabetes Mellitus; Hyperglycemia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- diabetes self-management education (Experimental): Diabetes survival skills self-management education (DSME) program content was aligned with American Diabetes Association and Joint Commission suggested key areas for hospital diabetes education. Content areas were as follows: when and how to take diabetes medications; glycemic goals and self-blood glucose monitoring; definition, prevention, recognition, and treatment of hypoglycemia and hyperglycemia; what to do before you see the dietitian; sick day management; and when to call the doctor or go to the ED. Program content was created for delivery via either DVD or print format.
  Interventions: Behavioral: diabetes self-management education

INTERVENTIONS:
Behavioral: diabetes self-management education — 1-group, pre-test/post-test design feasibility and preliminary efficacy evaluation of diabetes survival skills self-management education delivered at the hospital bedside.
  Other Names: survival skills education

SUMMARY:
A learner-centered diabetes survival skills self-management education program was provided to adults with uncontrolled diabetes in the hospital and generated preliminary evidence of impact on medication adherence and a trend toward reduction in hospital and emergency department admissions.

DETAILED DESCRIPTION:
This study was a prospective, nonrandomized pilot study conducted among adults with uncontrolled diabetes admitted to the Medicine Service of an urban tertiary teaching hospital were consented to participate in a pilot study which provided diabetes survival skills education. Based on knowledge deficits identified on a diabetes knowledge pre-test the patient was directed to view video content corresponding to those deficiencies and content on sick days and diabetes complications. Evaluation measures were diabetes knowledge, medication adherence, and hospital admissions plus emergency department visits at and/or 3months before baseline and at 2 weeks and 3 months post-discharge. There was improvement in diabetes knowledge and medication adherence, which was sustained to 3 months. A trend was observed toward reduction in emergency department and/or hospital admissions from 3 months pre-intervention to 3 months post-discharge for uncontrolled diabetes. This knowledge-based program successfully provided survival skills education to hospital patients with uncontrolled diabetes and demonstrated preliminary evidence of a positive impact on medication adherence and a trend toward reduction in hospital and emergency department admissions.

ELIGIBILITY:
Inclusion Criteria:

* English speaking with a diabetes mellitus diagnosis (ICD 9 codes 250.xx)
* an admitting blood glucose level of > 200 mg/dL or ≤ 40 mg/dL, and
* an anticipated hospital stay of ≥ 2 days, as estimated by the medical staff, to allow sufficient time for delivery of program content

Exclusion Criteria:

* pregnancy
* admission to an intensive care unit, and
* any medical condition or cognitive dysfunction that, in the opinion of the investigator, would preclude active participation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 125 (Actual)
Dates: Start 2010-05; Primary Completion 2011-11 (Actual); Study Completion 2011-11 (Actual)

PRIMARY OUTCOMES:
Assessment of change in Diabetes knowledge as measured by an 11-item diabetes knowledge survey | Baseline score obtained before receiving the education intervention. Post test score obtained immediately after the education intervention was completed during the hospital stay, usually within 24 hours or less from the baseline score
  11-item diabetes knowledge survey administered pre- and post- education intervention during the same hospital stay. Baseline score and post intervention score obtained within a 24 hour period

SECONDARY OUTCOMES:
Readmissions to the hospital and the emergency department | 3 months pre- and 3 months post-intervention
  Self-reported historic and post-intervention visits to ED and or admissions to the hospital
Medication adherence (Modified Morisky Medication Adherence Scale 4-item) | Baseline pre intervention then at 2 weeks after intervention and at 3 months post-intervention
  Modified Morisky Medication Adherence Scale 4-item

CONTACTS AND LOCATIONS:
Overall Officials: michelle f magee, MD, MBBCh,, Principal Investigator — Medstar Health Research Institute

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Magee MF, Khan NH, Desale S, Nassar CM. Diabetes to Go: Knowledge- and Competency-Based Hospital Survival Skills Diabetes Education Program Improves Postdischarge Medication Adherence. Diabetes Educ. 2014 May;40(3):344-350. doi: 10.1177/0145721714523684. Epub 2014 Feb 20. PMID 24557596

DOCUMENTS (1):
  • Informed Consent Form (2016-01-27): https://cdn.clinicaltrials.gov/large-docs/28/NCT03023228/ICF_000.pdf